CLINICAL TRIAL: NCT05804981
Title: Using the PROMIS Cognition Item Bank for Early Detection of Cognitive Decline in Primary Care
Brief Title: Early Detection of Cognitive Decline
Acronym: EDCD
Status: Withdrawn | Type: Observational
Why Stopped: study design revised and no longer fits definition of a clinical trial
Sponsor: RAND (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Pittsburgh Medical Center (Other); Northwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: HCQMI065; 5R61AG069776-02 (NIH)
Record Dates: First submitted 2022-09-30; First posted 2023-04-07 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Impairment
Keywords: cognitive decline; self-reported cognitive screener; annual wellness visit
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- new screener group: patients completing annual wellness visits after the new screener is adopted by the UPMC health system
  Interventions: Other: PRO-CS
- pre screener group: patients completing annual wellness visits before the new screener is adopted by the UPMC health system

INTERVENTIONS:
Other: PRO-CS — 4 questions about cognitive function added to annual wellness visit protocol
  Groups: new screener group

SUMMARY:
The goal of this clinical trial is to evaluate the impact of a brief cognitive screener on provider behavior in patients completing an annual wellness visit (AWV). The main question[s] it aims to answer are:

* do appropriate referrals increase for patients using the new screener?
* do appropriate diagnostic orders increase for patients using the new screener? Participants will respond to 4 questions about their cognitive abilities as part of a larger AWV protocol.

Researchers will compare provider behavior for patients completing AWVs before and after implementation of the new screener to see if referral, diagnostic and prescribing behaviors differ.

DETAILED DESCRIPTION:
In the course of this two-year project, the RAND team and partners (University of Pittsburgh Medical Center [UPMC] and Northwestern University [NU]) will conduct secondary data analysis to establish the validity of scores from the PCF item bank; use the resulting data to derive meaningful scoring criteria and interpretation guidance, and determine the best short form item set from the PCF item bank to use for standardized cognitive impairment screening during the Medicare Annual Wellness Visit (AWV); use qualitative methods to refine workflow for administering the screener in primary care; work with UPMC to integrate the resultant brief self-reported PROMIS cognition screener (PRO-CS) into their workflows; and evaluate the effect of implementing brief standardized PRO-CS with interpretive guidance on primary care providers' behaviors. The control group will consist of all digital records of annual wellness visits in the year prior to implementation of the PRO-CS

ELIGIBILITY:
Inclusion Criteria:

* has AWV within study period

Exclusion Criteria:

* provider uses non-digital AWV form

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: all patients aged 65 and older who completed annual wellness visits within the study period at participating clinics within the UPMC system
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-01-19 (Estimated); Study Completion 2024-01-19 (Estimated)

PRIMARY OUTCOMES:
specialist referrals | within one month post AWV
  referrals to specialists for cognitive impairment (e.g., neurology, social work, geriatrics) as found in patient EMR. Specialist referrals include neurology, neuropsychology, psychiatry, psychology, social worker, geriatrics.
diagnostic orders | within one month post AWV
  diagnostic orders to rule out reversible causes of CI as found in patient EMR. Orders include those for TSH, B12, RPR, or head imaging

CONTACTS AND LOCATIONS:
Overall Officials: Maria Edelen, PhD, Principal Investigator — RAND
Locations (1):
- University of Pittsburg Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No